CLINICAL TRIAL: NCT00803374
Title: A Phase I, Multiple Ascending Dose Study of BMS-663513 (Anti CD137) in Combination With Ipilimumab (BMS-734016/Anti-CTLA-4) in Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: Combination of Anti-CD137 & Ipilimumab in Patients With Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA186-007
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — urelumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.1 mg/kg (Experimental)
  Interventions: Drug: AntiCD137; Drug: Ipilimumab
- 0.3 mg/kg (Experimental)
  Interventions: Drug: AntiCD137; Drug: Ipilimumab
- 1.0 mg/kg (Experimental)
  Interventions: Drug: AntiCD137; Drug: Ipilimumab
- 3.0 mg/kg (Experimental)
  Interventions: Drug: AntiCD137; Drug: Ipilimumab
- 10 mg/kg (Experimental)
  Interventions: Drug: AntiCD137; Drug: Ipilimumab

INTERVENTIONS:
Drug: AntiCD137 — Infusion, IV, 0.1 mg/kg, Q3 weeks for 12 weeks then Q12 weeks, 12+ weeks depending on response
  Other Names: BMS-663513
  Arms: 0.1 mg/kg
Drug: AntiCD137 — Infusion, IV, 0.3 mg/kg, Q3 weeks for 12 weeks then Q12 weeks, 12+ weeks depending on response
  Other Names: BMS-663513
  Arms: 0.3 mg/kg
Drug: AntiCD137 — Infusion, IV, 1.0 mg/kg, Q3 weeks for 12 weeks then Q12 weeks, 12+ weeks depending on response
  Other Names: BMS-663513
  Arms: 1.0 mg/kg
Drug: AntiCD137 — Infusion, IV, 3.0 mg/kg, Q3 weeks for 12 weeks then Q12 weeks, 12+ weeks depending on response
  Other Names: BMS-663513
  Arms: 3.0 mg/kg
Drug: AntiCD137 — Infusion, IV, 10 mg/kg, Q3 weeks for 12 weeks then Q12 weeks, 12+ weeks depending on response
  Other Names: BMS-663513
  Arms: 10 mg/kg
Drug: Ipilimumab — Infusion, IV, 10 mg/kg, Q3 weeks for 12 weeks then Q12, 12+ weeks depending on response
  Other Names: BMS-734016; MDX-010

SUMMARY:
The purpose of this study is to determine if BMS-663513 administered in combination with ipilimumab to patients with advanced malignant melanoma is safe and tolerable

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant melanoma
* Stage III (unresectable) or Stage IV disease which may have been treated with up to one prior cytotoxic chemotherapy and/or up to 3 other therapeutic regimens
* Willing to undergo up to 3 biopsies of an accessible lesion

Exclusion Criteria:

* Active/symptomatic brain metastases
* Primary ocular melanoma or primary tumor of unknown origin
* Concurrent autoimmune disease
* Previous treatment with a CD137 agonist or CTLA-4 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of safety and tolerability as determined by analysis of adverse event reports and results of vital sign measurements, physical examinations, and clinical laboratory tests | During the course of the each subject's treatment and up to 70 days after his or her last dose of study medication is received

SECONDARY OUTCOMES:
Evidence of clinical improvement in tumor burden confirmed by CT or MRI | Weeks 12, 18, 24, 30, 36, 42, 48, and every 12 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Local Institution, Los Angeles, California
  - Local Institution, New Haven, Connecticut
  - Local Institution, Tampa, Florida
  - Local Institution, Boston, Massachusetts
  - Local Institution, New York, New York

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx